CLINICAL TRIAL: NCT05659082
Title: Cognition and Magnetic Resonance Imaging After Psychiatric Neurosurgery for Intractable Obsessive-Compulsive Disorder- Phase 2
Brief Title: Ventral Capsulotomy for Intractable OCD
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Nicole McLaughlin, Research Psychologist, Associate Professor, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1909-001
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Laser Interstitial Thermal Therapy — Ventral capsulotomy for OCD using laser interstitial thermal therapy

SUMMARY:
Obsessive-compulsive disorder impacts 1-2 percent of the population. Unfortunately, about fifteen percent of patients fail to benefit from existing therapies. A small number of OCD patients, who have a disabling illness that does not improve after conventional treatments, have neurosurgery as a last resort. One procedure, capsulotomy, involves making pairs of lesions in an anatomically-defined part of the anterior limb of the internal capsule, a structure containing nerve fiber bundles connecting the thalamus, in the center of the brain, to the prefrontal cortex, the most anterior and outermost brain region. The investigators will examine how the therapeutic effects of capsulotomy relate to changes in the structure of these brain pathways with structural (diffusion tensor imaging, DTI) and functional (resting-state and task-based) connectivity metrics. The investigators will also utilize experimental cognitive tasks that are sensitive to the circuitry impacted by this procedure.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a common condition. One to two percent of the population experiences the chronic intrusive obsessive thoughts, repetitive compulsions, and pathological anxiety characteristic of the illness, which by several measures is among the ten most disabling medical conditions for adults in industrialized countries. Unfortunately, about fifteen percent of patients fail to benefit from existing therapies. A small number of OCD patients, who have a disabling illness that does not improve after conventional treatments, have neurosurgery as a last resort. One procedure, capsulotomy, involves making pairs of lesions in an anatomically-defined part of the anterior limb of the internal capsule, a structure containing nerve fiber bundles connecting the thalamus, in the center of the brain, to the prefrontal cortex, the most anterior and outermost brain region. OCD is believed to result from abnormal activity in brain circuits connecting the prefrontal cortex, thalamus and other brain areas. Data show that approximately 50 to 60 percent of patients improve after capsulotomy.

In addition, new neuroimaging measures of how brain fiber tracts and the brain regions associated with them change after capsulotomy promise to enhance the understanding of OCD pathophysiology, and may help advance capsulotomy and other neuroanatomically-based therapies. While capsulotomy is believed to exert its therapeutics effects by changing thalamus-prefrontal cortex connections, the specific anatomical changes produced by this surgical treatment in these fiber pathways are unknown. This is especially true at greater distances from the site of surgery, that is, closer to the thalamus and prefrontal cortex, the regions the surgery is intended to partially disconnect from each other. The investigators will examine how the therapeutic effects of capsulotomy relate to changes in the structure of these brain pathways with structural (diffusion tensor imaging, DTI) and functional (resting-state and task-based) connectivity metrics. Additional measures of how brain volumes may change in specific corticobasal structures implicated in OCD (including the basal ganglia, thalamus, and orbitofrontal cortex) will be derived from conventional MRI measures obtained during the same sessions when the experimental DT-MRI measures are acquired. The investigators will also utilize experimental cognitive tasks that are sensitive to the circuitry impacted by this procedure.

Understanding the changes after surgery that result in the best therapeutic outcomes will allow the investigators to improve capsulotomy as a treatment for this debilitating disease. With this information, the investigators can refine the targeting of capsulotomy for individual patients and, possibly, aid the development of other treatments, including deep brain stimulation, for intractable OCD. This study provides a unique opportunity to test structural and functional connectivity measures as probes of complex neuronal circuits that are likely to be involved in psychiatric illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be undergoing capsulotomy for severe OCD, as approved by the Butler Hospital Psychiatric Neurosurgery Committee

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 12 months
  Change from baseline to 12 months on YBOCS score; YBOCS score ranges from 0-40, and higher scores indicate more severe illness
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 24 months
  Change from baseline to 24 months on YBOCS score; YBOCS score ranges from 0-40, and higher scores indicate more severe illness

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | 12 months
  Change from baseline to 12 months on HDRS score; HRDS scores range from 0-52, with higher scores indicating more severe illness
Hamilton Anxiety Rating Scale (HARS) | 12 months
  Change from baseline to 12 months on HARS score; HARS score ranges from 0-56, with higher scores indicating more severe illness

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided